CLINICAL TRIAL: NCT00649545
Title: A Multi-Center Study of the Safety and Efficacy of Human Anti-TNF Monoclonal Antibody Adalimumab (D2E7) in Patients With Active Rheumatoid Arthritis
Brief Title: Study of the Human Anti-TNF Monoclonal Antibody in Patients With Active Rheumatoid Arthritis
Acronym: CanAct
Status: Approved for marketing | Type: Expanded Access
Sponsor: Abbott (Industry)
Responsible Party: Larry McNamee, Sr. clinical Research Manager, Abbott
Other Study IDs: M02-574
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

INTERVENTIONS:
Biological: adalimumab — 40 mg every other week
  Other Names: ABT-D2E7; Humira

SUMMARY:
The primary objective of this study is to assess the safety (by collecting adverse events and serious adverse events) of adalimumab administered every other week to patients with moderately to severly active rheumatoid arthritis who have failed prior disease-modifying anti-rheumatic drugs (DMARDs).

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed (i.e. not dropped out of) the DE013 study or fulfills criteria 2-12
* Patients 18 years of age or older
* Female is either not childbearing, defined as post-menopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or if childbearing potential, practicing an acceptable method of birth control
* Female of childbearing potential must have a negative serum pregnancy test prior to first dose of adalimumab
* Diagnosis of active RA defined by >= 5 swollen joints and one of the following:

  * Positive RF
  * One or more joint erosions present of x-ray
  * HAQ score > 1

Exclusion Criteria:

* Patient has failed 2 or more biologics
* Patient who had previous treatment with cyclophosphamide and chlorambucil
* Previous treatment with total lymphoid irradiation or anti-CD4 or CAMPATH 1H monoclonal antibody resulting in presistent CD4 lymphopenia (CD4 lymphocytes +< 500/mm3)
* History of cancer within the past 10 years unless successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix
* History of malignant lymphoma or leukemia regardless of treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778
- [Derived] Haraoui B, Cividino A, Stewart J, Guerette B, Keystone EC. Safety and effectiveness of adalimumab in a clinical setting that reflects Canadian standard of care for the treatment of rheumatoid arthritis (RA): results from the CanACT study. BMC Musculoskelet Disord. 2011 Nov 17;12:261. doi: 10.1186/1471-2474-12-261. PMID 22093579